CLINICAL TRIAL: NCT04424550
Title: Comparative Long-term Results After DSAEK, UT-DSAEK and DMEK for Fuchs Endothelial Corneal Dystophy and Moderated Pseudophakic Bullous Keratopathy
Brief Title: Comparative Results After DSAEK, UT-DSAEK and DMEK for Fuchs Endothelial Corneal Dystophy
Acronym: DEMOGRAFT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-01Obs-CHRMT
Record Dates: First submitted 2020-06-03; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Corneal Dystrophy
Keywords: DMEK, DSAEK, UT-DSAEK, Endothelial cell
MeSH Terms: conditions — Corneal Dystrophies, Hereditary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Purpose of the research is to describe and compare the evolution of BSCVA after DMEK, DSAEK and UT-DSAEK for Fuchs Endothelial Corneal Dystrophy (FECD) and Moderate Pseudophakic Bullous Keratopathy (PBK). To secondarily research the correlates criterions with best spectacle corrected visual acuity (BSCVA) 12 months postoperatively.

DETAILED DESCRIPTION:
The purpose of the research is to Describe and compare the evolution of BSCVA after DMEK, DSAEK and UT-DSAEK for Fuchs Endothelial Corneal Dystrophy (FECD) and Moderate Pseudophakic Bullous Keratopathy (PBK). To secondarily research the correlates criterions with best spectacle corrected visual acuity (BSCVA) 12 months postoperatively.

In a retrospective, single-center, observational study, 218 eyes treated with DMEK (n=110), UT-DSAEK (n=58) and DSAEK (n=50) surgeries were studied. Patients requiring posterior lamellar transplantation for FECD or moderate PBK, with preoperative BSCVA of less than 0.3 logmar, were selected. Patients with pathologies that may seriously affect VA postoperatively were excluded. Graft thickness for DSAEK was measured during the surgery and in vivo at D8, D15, M1, M6, M12 and M24. The primary endpoint was best spectacle corrected visual acuity (BSCVA) in logMAR at 6, 12 and 24 months. We deliberately differentiated our postoperative visual results by comparing DMEK with DSAEK or UT-DSAEK with central graft thickness (CGT) measurements carried out either pre-operatively (less than or greater than 130 µm) or post-operatively at 6 months (less than or greater than 100µm). Type of endothelial graft, Donor and recipient's ages, Graft's endothelial cell density (ECD), Rebubbling rate, preoperative VA, graft's indications and surgical time were also tested to explain BSCVA at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring posterior lamellar transplantation for FECD or moderate PBK, with preoperative BSCVA of less than 0.3 logmar,

Exclusion Criteria:

* Patients with pathologies that may seriously affect VA postoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study included patients who had undergone posterior lamellar keratoplasty for FECD or moderate PBK indications with a minimum follow-up period of 24 months. The surgical procedures were either DMEK, DSAEK or UT-DSAEK and were performed by the same experienced surgeon (JMP).
Sampling Method: Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
visual acuity | 6 months
  The primary endpoint was best spectacle corrected visual acuity (BSCVA) in logMAR at 6 months
visual acuity | 12 months
  The primary endpoint was best spectacle corrected visual acuity (BSCVA) in logMAR at 12 months
visual acuity | 24 months
  The primary endpoint was best spectacle corrected visual acuity (BSCVA) in logMAR at 24 months

SECONDARY OUTCOMES:
central graft thickness measurements | 6 months
  central graft thickness (CGT) measurements carried out either pre-operatively (less than or greater than 130 µm) or post-operatively at 6 months (less than or greater than 100µm)
Type of endothelial graft | days 1
  Type of endothelial graft
Donor's ages | days 1
  Donor's ages
recipient's ages | day 1
  recipient's ages
Graft's endothelial cell density | day 1
  Graft's endothelial cell density was evaluated via no-contact specular microscopy (NIDEK CEM-530 NIDEK CO. LTD).
Rebubbling rate | day 1
  Rebubbling rate
Preoperative visual acuity | day 1
  Preoperative visual acuity was scored with reference to the logarithm of the minimum angle of resolution (LogMAR).
graft's indications | day 1
  The indications of the grafts are different between the DMEK groups and the DSAEK and or UT-DSAEK groups: Fuchs endothelial corneal dystrophies (FECD) and moderated pseudophakic bullous keratopathies (PBK)
surgical time | day 1
  surgical time

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc PERONE, MD, Principal Investigator — CHR Metz Thionville
Locations (1):
- Chr Metz Thionville, Metz, France

REFERENCES:
- [Derived] Perone JM, Goetz C, Zevering Y, Derumigny A. Principal Component Analysis of a Real-World Cohort of Descemet Stripping Automated Endothelial Keratoplasty and Descemet Membrane Endothelial Keratoplasty Cases: Demonstration of a Powerful Data-Mining Technique for Identifying Areas of Research. Cornea. 2025 Feb 1;44(2):209-220. doi: 10.1097/ICO.0000000000003584. Epub 2024 May 29. PMID 38830189
- [Derived] Perone JM, Goetz C, Zevering Y, Derumigny A, Bloch F, Vermion JC, Lhuillier L. Graft Thickness at 6 Months Postoperatively Predicts Long-Term Visual Acuity Outcomes of Descemet Stripping Automated Endothelial Keratoplasty for Fuchs Dystrophy and Moderate Phakic Bullous Keratopathy: A Cohort Study. Cornea. 2022 Nov 1;41(11):1362-1371. doi: 10.1097/ICO.0000000000002872. Epub 2021 Oct 22. PMID 34690269